CLINICAL TRIAL: NCT02593786
Title: A Phase 1/2, Open-Label Study of Nivolumab (BMS-936558) in Chinese Subjects With Previously Treated Advanced or Recurrent Solid Tumors (CheckMate 077: CHECKpoint Pathway and nivoluMAb Clinical Trial Evaluation 077)
Brief Title: A Study of Safety, Tolerability and Pharmacokinetics of Nivolumab in Chinese Subjects With Previously Treated Advanced or Recurrent Solid Tumors
Acronym: CheckMate 077
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-077
Record Dates: First submitted 2015-10-30; First posted 2015-11-02 (Estimated); Results first posted 2022-10-24 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-09

CONDITIONS: Solid Tumors
MeSH Terms: interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Nivolumab monotherapy (Experimental): Nivolumab specified dose on specified days
  Interventions: Drug: Nivolumab
- Cohort Expansion (Experimental): Nivolumab specified dose on specified days
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab

SUMMARY:
The purpose of this study is to determine whether nivolumab is safe and effective in the treatment of advanced or recurrent solid tumors in Chinese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Chinese subjects with advanced or recurrent solid tumors

Exclusion Criteria:

* Subjects with brain metastases are excluded unless clinically stable for more than 2 weeks at the time of enrollment as determined by the investigator
* Subjects with carcinomatous meningitis are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2016-01-07 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2021-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- China (2):
  - Local Institution - 0001, Guangzhou, Guangdong
  - Local Institution, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Ma Y, Fang W, Zhang Y, Yang Y, Hong S, Zhao Y, Tendolkar A, Chen L, Xu D, Sheng J, Zhao H, Zhang L. A Phase I/II Open-Label Study of Nivolumab in Previously Treated Advanced or Recurrent Nasopharyngeal Carcinoma and Other Solid Tumors. Oncologist. 2019 Jul;24(7):891-e431. doi: 10.1634/theoncologist.2019-0284. Epub 2019 May 2. PMID 31048330
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A: Nivolumab 3 mg/kg Q2W: Participants receive nivolumab (3 mg/kg) administered as 4 doses in each 8-week treatment cycle at Days 1, 15, 29 and 43.
- Cohort B: Nivolumab 240 mg Q2W: Participants receive a flat dose of nivolumab (240 mg) administered as 4 doses in each 8-week treatment cycle at Days 1, 15, 29 and 43.
- Cohort C: Nivolumab 360 mg Q3W: Participants receive a flat dose of nivolumab (360 mg) administered as one dose in each 3-week treatment cycle.
- Cohort D: Nivolumab 480 mg Q4W: Participants receive a flat dose of nivolumab (480 mg) administered as one dose in each 4-week treatment cycle
Period: Overall Study
Arm/Group | Cohort A: Nivolumab 3 mg/kg Q2W | Cohort B: Nivolumab 240 mg Q2W | Cohort C: Nivolumab 360 mg Q3W | Cohort D: Nivolumab 480 mg Q4W
Started | 15 | 20 | 11 | 12
Completed | 0 | 0 | 0 | 0
Not Completed | 15 | 20 | 11 | 12
Not completed — Disease progression | 12 | 16 | 10 | 7
Not completed — Study drug toxicity | 1 | 0 | 0 | 0
Not completed — Adverse event unrelated to study drug | 1 | 1 | 1 | 0
Not completed — Participant request to discontinue study therapy | 0 | 2 | 0 | 0
Not completed — Other reasons | 1 | 1 | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: Nivolumab 3 mg/kg Q2W | Cohort B: Nivolumab 240 mg Q2W | Cohort C: Nivolumab 360 mg Q3W | Cohort D: Nivolumab 480 mg Q4W | Total
Number analyzed (Participants) | 15 | 20 | 11 | 12 | 58
Age, Customized [Count of Participants; unit: Participants]
  > 65 | 15 | 20 | 10 | 9 | 54
  >= 65 | 0 | 0 | 1 | 3 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 4 | 5 | 20
  Male | 11 | 13 | 7 | 7 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 15 | 20 | 11 | 12 | 58
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants Experiencing Drug-Related Grade 3-4 Adverse Events (AEs)
Description: A drug related adverse event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study drug that has a causal relationship with the treatment. AEs are graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (Version 4.03) (NCI CTCAE) guidelines where Grade 3= Severe and Grade 4= Life-threatening.
Time Frame: From first dose to 100 days after last dose (up to approximately 28 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Nivolumab 3 mg/kg Q2W | Cohort B: Nivolumab 240 mg Q2W | Cohort C: Nivolumab 360 mg Q3W | Cohort D: Nivolumab 480 mg Q4W
Number analyzed (Participants) | 15 | 20 | 11 | 12
Participants | 1 | 1 | 0 | 0

2. Primary Outcome: The Number of Participants Experiencing Drug-Related Grade 3-4 Serious Adverse Events (SAEs)
Description: A drug related serious adverse event (SAE) is any untoward medical occurrence that at any dose: results in death; is life-threatening; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; or is an important medical event that has a casual relationship with the treatment. SAEs are graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (Version 4.03) (NCI CTCAE) guidelines where Grade 3= Severe and Grade 4= Life-threatening.
Time Frame: From first dose to 100 days after last dose (up to approximately 28 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Groups:
- Cohort C: Nivolumab 360 mg Q3W: Participants receive a flat dose of nivolumab (360 mg) in each 3-week treatment cycle.
- Cohort D: Nivolumab 480 mg Q4W: Participants receive a flat dose of nivolumab (480 mg) in each 4-week treatment cycle
Arm/Group | Cohort A: Nivolumab 3 mg/kg Q2W | Cohort B: Nivolumab 240 mg Q2W | Cohort C: Nivolumab 360 mg Q3W | Cohort D: Nivolumab 480 mg Q4W
Number analyzed (Participants) | 15 | 20 | 11 | 12
Participants | 0 | 1 | 0 | 0

3. Primary Outcome: The Number of Participants Experiencing Abnormal Hepatic Laboratory Test Results
Description: The number of participants with the following laboratory abnormalities from the following on-treatment evaluations:
  * ALT or AST > 3 x ULN, > 5 x ULN, > 10 x ULN and > 20 x ULN
  * Total bilirubin > 2 x ULN
  * Concurrent (within 1 day) ALT or AST > 3 x ULN and total bilirubin > 2 x ULN
  * Concurrent (within 30 days) ALT or AST > 3 x ULN and total bilirubin > 2 x ULN
Time Frame: From first dose to 100 days after last dose (up to approximately 28 months)
Population: All treated participants with least one on-treatment measurement of the corresponding laboratory parameter
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Nivolumab 3 mg/kg Q2W | Cohort B: Nivolumab 240 mg Q2W | Cohort C: Nivolumab 360 mg Q3W | Cohort D: Nivolumab 480 mg Q4W
Number analyzed (Participants) | 13 | 20 | 10 | 12
Participants
  ALT OR AST > 3XULN | 0 | 3 | 0 | 1
  ALT OR AST> 5XULN | 0 | 2 | 0 | 0
  ALT OR AST> 10XULN | 0 | 1 | 0 | 0
  ALT OR AST > 20XULN | 0 | 0 | 0 | 0
  TOTAL BILIRUBIN > 2XULN | 0 | 3 | 1 | 0
  ALT/AST ELEV>3XULN;TOTAL BILIRUBIN>2XULN IN 1 DAY | 0 | 3 | 0 | 0
  ALT/AST ELEV>3XULN;TOTAL BILIRUBIN>2XULN IN 30 DAYS | 0 | 3 | 0 | 0

4. Secondary Outcome: Best Overall Response (BOR)
Description: Best overall response (BOR) was assessed by the investigator using Response Evaluation Criteria in Solid Tumor (RECIST v1.1). Complete Response (CR) is defined as a disappearance of all target lesions. Partial Response (PR) is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Stable Disease (SD) is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. Progressive Disease (PD) is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study).
Time Frame: From first dose up to approximately 28 months
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Nivolumab 3 mg/kg Q2W | Cohort B: Nivolumab 240 mg Q2W | Cohort C: Nivolumab 360 mg Q3W | Cohort D: Nivolumab 480 mg Q4W
Number analyzed (Participants) | 15 | 20 | 11 | 12
Participants
  Complete Response | 0 | 0 | 0 | 0
  Partial Response | 3 | 2 | 1 | 2
  Stable Disease | 2 | 12 | 6 | 6
  Progressive Disease | 9 | 5 | 4 | 4
  Unable to Determine | 1 | 1 | 0 | 0

5. Secondary Outcome: Duration of Response (DOR)
Description: Duration of response is defined as the time from the date of first response (CR or PR) to the date of the first documented tumor progression as determined using RECIST 1.1 or death due to any cause, whichever occurs first. Participants who remain alive and have not progressed will be censored on the date of their last tumor assessment. Participants who started subsequent therapy without a prior reported progression will be censored at the last tumor assessment prior to initiation of the subsequent anticancer therapy. Complete response (CR) is defined as a disappearance of all target lesions and partial response (PR) is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Other tumor types include: gastric, melanoma, neuroblastoma, colorectal cancer, cervical cancer, duodenal papillary carcinoma, and gallbladder carcinoma.
Time Frame: From the date of first response (CR or PR) to the date of the first documented tumor progression or death due to any cause, whichever occurs first. (Up to approximately 28 months)
Population: All treated participants with a BOR of CR or PR
Measure: Median (Full Range); unit: Weeks
Arm/Group | Cohort A: Nivolumab 3 mg/kg Q2W | Cohort B: Nivolumab 240 mg Q2W | Cohort C: Nivolumab 360 mg Q3W | Cohort D: Nivolumab 480 mg Q4W
Number analyzed (Participants) | 3 | 2 | 1 | 2
Weeks
  Hepatocellular carcinoma: number analyzed (Participants) | 0 | 0 | 0 | 1
  Hepatocellular carcinoma |  |  |  | NA [95.3 to 95.3] — Insufficient number of participants with events
  Non-small cell lung carcinoma (NSCLC): number analyzed (Participants) | 1 | 0 | 1 | 0
  Non-small cell lung carcinoma (NSCLC) | NA [8.3 to 8.3] — Insufficient number of participants with events |  | 6.1 [6.1 to 6.1] |
  Nasopharyngeal carcinoma: number analyzed (Participants) | 2 | 2 | 0 | 1
  Nasopharyngeal carcinoma | NA [48.7 to 75.7] — Insufficient number of participants with events | NA [34.1 to 81.1] — Insufficient number of participants with events |  | NA [83.3 to 83.3] — Insufficient number of participants with events
  Other tumor types: number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Objective Response Rate (ORR)
Description: Objective response rate (ORR) is defined as the percentage of all treated participants whose best overall response (BOR) is either a complete response (CR) or partial response (PR) by investigator using Response Evaluation Criteria in Solid Tumor (RECIST v1.1). Complete response (CR) is defined as a disappearance of all target lesions and partial response (PR) is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Other tumor types include: gastric, melanoma, neuroblastoma, colorectal cancer, cervical cancer, duodenal papillary carcinoma, and gallbladder carcinoma.
Time Frame: From first dose up to approximately 28 months
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Cohort A: Nivolumab 3 mg/kg Q2W | Cohort B: Nivolumab 240 mg Q2W | Cohort C: Nivolumab 360 mg Q3W | Cohort D: Nivolumab 480 mg Q4W
Number analyzed (Participants) | 15 | 20 | 11 | 12
Percent of participants
  Hepatocellular carcinoma: number analyzed (Participants) | 0 | 2 | 0 | 1
  Hepatocellular carcinoma |  | 0 [NA to NA] — Insufficient number of participants with events |  | 100 [NA to NA] — Insufficient number of participants with events
  Non-small cell lung carcinoma (NSCLC): number analyzed (Participants) | 9 | 1 | 1 | 3
  Non-small cell lung carcinoma (NSCLC) | 11.1 [NA to NA] — Insufficient number of participants with events | 0 [NA to NA] — Insufficient number of participants with events | 100 [NA to NA] — Insufficient number of participants with events | 0 [NA to NA] — Insufficient number of participants with events
  Nasopharyngeal carcinoma: number analyzed (Participants) | 6 | 17 | 10 | 1
  Nasopharyngeal carcinoma | 33.3 [NA to NA] — Insufficient number of participants with events | 11.8 [1.5 to 36.4] | 0 [0.0 to 30.8] | 100 [NA to NA] — Insufficient number of participants with events
  Other tumor types: number analyzed (Participants) | 0 | 0 | 0 | 7
  Other tumor types |  |  |  | 0 [NA to NA] — Insufficient number of participants with events

7. Secondary Outcome: Response Rate at 24 Weeks
Description: Response rate at 24 weeks is defined as the percentage of all treated participants who have CR or PR by 24 weeks. Complete response (CR) is defined as a disappearance of all target lesions and partial response (PR) is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Other tumor types include: gastric, melanoma, neuroblastoma, colorectal cancer, cervical cancer, duodenal papillary carcinoma, and gallbladder carcinoma.
Time Frame: Week 24
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Cohort A: Nivolumab 3 mg/kg Q2W | Cohort B: Nivolumab 240 mg Q2W | Cohort C: Nivolumab 360 mg Q3W | Cohort D: Nivolumab 480 mg Q4W
Number analyzed (Participants) | 15 | 20 | 11 | 12
Percent of participants
  Hepatocellular carcinoma: number analyzed (Participants) | 0 | 2 | 0 | 1
  Hepatocellular carcinoma |  | 0 [NA to NA] — Insufficient number of participants with events |  | 100 [NA to NA] — Insufficient number of participants with events
  Non-small cell lung carcinoma (NSCLC): number analyzed (Participants) | 9 | 1 | 1 | 3
  Non-small cell lung carcinoma (NSCLC) | 11.1 [NA to NA] — Insufficient number of participants with events | 0 [NA to NA] — Insufficient number of participants with events | 100 [NA to NA] — Insufficient number of participants with events | 0 [NA to NA] — Insufficient number of participants with events
  Nasopharyngeal carcinoma: number analyzed (Participants) | 6 | 17 | 10 | 1
  Nasopharyngeal carcinoma | 33.3 [NA to NA] — Insufficient number of participants with events | 5.9 [0.1 to 28.7] | 0 [0.0 to 30.8] | 100 [NA to NA] — Insufficient number of participants with events
  Other tumor types: number analyzed (Participants) | 0 | 0 | 0 | 7
  Other tumor types |  |  |  | 0 [NA to NA] — Insufficient number of participants with events

8. Secondary Outcome: Disease Control Rate (DCR) at 24 Weeks
Description: Disease control rate (DCR) at 24 weeks is defined as the percentage of all treated participants who have CR, PR or SD by 24 weeks. Complete Response (CR) is defined as a disappearance of all target lesions. Partial Response (PR) is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Stable Disease (SD) is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. Other tumor types include: gastric, melanoma, neuroblastoma, cervical cancer, duodenal papillary carcinoma, and gallbladder carcinoma.
Time Frame: Week 24
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Cohort A: Nivolumab 3 mg/kg Q2W | Cohort B: Nivolumab 240 mg Q2W | Cohort C: Nivolumab 360 mg Q3W | Cohort D: Nivolumab 480 mg Q4W
Number analyzed (Participants) | 15 | 20 | 11 | 12
Percent of participants
  Colorectal Cancer: number analyzed (Participants) | 0 | 0 | 0 | 1
  Colorectal Cancer |  |  |  | 100 [NA to NA] — Insufficient number of participants with events
  Hepatocellular carcinoma: number analyzed (Participants) | 0 | 2 | 0 | 1
  Hepatocellular carcinoma |  | 0 [NA to NA] — Insufficient number of participants with events |  | 100 [NA to NA] — Insufficient number of participants with events
  Non-small cell lung carcinoma (NSCLC): number analyzed (Participants) | 9 | 1 | 1 | 3
  Non-small cell lung carcinoma (NSCLC) | 11.1 [NA to NA] — Insufficient number of participants with events | 0 [NA to NA] — Insufficient number of participants with events | 100 [NA to NA] — Insufficient number of participants with events | 66.7 [NA to NA] — Insufficient number of participants with events
  Nasopharyngeal carcinoma: number analyzed (Participants) | 6 | 17 | 10 | 1
  Nasopharyngeal carcinoma | 33.3 [NA to NA] — Insufficient number of participants with events | 23.5 [6.8 to 49.9] | 20.0 [2.5 to 55.6] | 100 [NA to NA] — Insufficient number of participants with events
  Other tumor types: number analyzed (Participants) | 0 | 0 | 0 | 6
  Other tumor types |  |  |  | 0 [NA to NA] — Insufficient number of participants with events

9. Secondary Outcome: The Number of Participants With Positive Anti Drug Antibody (ADA) Assessments at Baseline and Positive or Negative ADA Samples After Treatment
Description: The number of participants with the following anti-drug responses:
  1. Baseline ADA positive: all participants with baseline ADA positive samples.
  2. ADA Positive: participants that have at least one ADA positive sample relative to baseline at any time after initiation of treatment.
  3. ADA negative: participants that have no ADA positive samples after the initiation of treatment.
Time Frame: From pre-dose on day 1 Cycle 1 up to participants end of study (up to approximately 28 months)
Population: All Nivolumab Treated Participants with Baseline and at Least One Post-baseline Assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Nivolumab 3 mg/kg Q2W | Cohort B: Nivolumab 240 mg Q2W | Cohort C: Nivolumab 360 mg Q3W | Cohort D: Nivolumab 480 mg Q4W
Number analyzed (Participants) | 13 | 19 | 10 | 12
Participants
  ADA positive sample at baseline | 1 | 4 | 0 | 0
  ADA positive sample after initiation of treatment | 1 | 0 | 0 | 2
  ADA Negative sample after initiation of treatment | 12 | 19 | 10 | 10

10. Secondary Outcome: Cmax - Maximum Observed Serum Concentration
Description: Nivolumab pharmacokinetic parameters are derived from serum concentration versus time data. Cmax is the maximum observed serum concentration over time.
Time Frame: Day 1 Cycle 1, 3, 5, 6 (pre-dose, 0.5, 4, 8, 24, 48, 96, 168, hours post dose. Cohort C-D includes also 336 hours post dose)
Population: All treated participants with evaluable serum concentration data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Cohort A: Nivolumab 3 mg/kg Q2W | Cohort B: Nivolumab 240 mg Q2W | Cohort C: Nivolumab 360 mg Q3W | Cohort D: Nivolumab 480 mg Q4W
Number analyzed (Participants) | 15 | 20 | 11 | 12
ug/mL
  Cycle 1 Day 1 | 57.025 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 18 | 77.674 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 18 | 108.455 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 21 | 206.630 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 22
  Cycle 3 Day 1: number analyzed (Participants) | 7 | 9 | 0 | 0
  Cycle 3 Day 1 | 132.222 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 17 | 171.604 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 14 |  |
  Cycle 5 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 6
  Cycle 5 Day 1 |  |  |  | 265.550 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 17
  Cycle 6 Day 1: number analyzed (Participants) | 0 | 0 | 7 | 0
  Cycle 6 Day 1 |  |  | 165.369 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 24 |

11. Secondary Outcome: Tmax - Time of Maximum Observed Serum Concentration
Description: Nivolumab pharmacokinetic parameters are derived from serum concentration versus time data. Tmax is the time of maximum observed serum concentration.
Time Frame: as for outcome 10
Population: All treated participants with evaluable serum concentration data
Measure: Median (Full Range); unit: h
Arm/Group | Cohort A: Nivolumab 3 mg/kg Q2W | Cohort B: Nivolumab 240 mg Q2W | Cohort C: Nivolumab 360 mg Q3W | Cohort D: Nivolumab 480 mg Q4W
Number analyzed (Participants) | 15 | 20 | 11 | 12
h
  Cycle 1 Day 1 | 4.00 [0.5 to 4.0] | 4.00 [0.5 to 8.0] | 4.0 [4.0 to 8.0] | 4.01 [0.5 to 8.0]
  Cycle 3 Day 1: number analyzed (Participants) | 7 | 9 | 0 | 0
  Cycle 3 Day 1 | 8.00 [4.0 to 48.2] | 8.00 [4.0 to 48.0] |  |
  Cycle 5 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 6
  Cycle 5 Day 1 |  |  |  | 2.26 [0.5 to 8.0]
  Cycle 6 Day 1: number analyzed (Participants) | 0 | 0 | 7 | 0
  Cycle 6 Day 1 |  |  | 8.00 [0.5 to 24.1] |

12. Secondary Outcome: AUC (0-T)-Area Under the Plasma Concentration-Time Curve
Description: Nivolumab pharmacokinetic parameters are derived from serum concentration versus time data. AUC (0-T) is the area under the plasma concentration-time curve from time zero to the last time of the last quantifiable concentration.
Time Frame: as for outcome 10
Population: All treated participants with evaluable serum concentration data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Cohort A: Nivolumab 3 mg/kg Q2W | Cohort B: Nivolumab 240 mg Q2W | Cohort C: Nivolumab 360 mg Q3W | Cohort D: Nivolumab 480 mg Q4W
Number analyzed (Participants) | 15 | 20 | 11 | 12
h*ug/mL
  Cycle 1 Day 1: number analyzed (Participants) | 15 | 20 | 10 | 12
  Cycle 1 Day 1 | 8353.429 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 29 | 11646.854 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 27 | 23567.315 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 17 | 49115.208 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 17
  Cycle 3 Day 1: number analyzed (Participants) | 7 | 9 | 0 | 0
  Cycle 3 Day 1 | 28442.153 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 28 | 35649.049 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 28 |  |
  Cycle 5 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 6
  Cycle 5 Day 1 |  |  |  | 91967.438 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 35
  Cycle 6 Day 1: number analyzed (Participants) | 0 | 0 | 7 | 0
  Cycle 6 Day 1 |  |  | 51087.588 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 44 |

13. Secondary Outcome: AUC(TAU) - Area Under the Concentration-Time Curve in One Dosing Interval
Description: Nivolumab pharmacokinetic parameters are derived from serum concentration versus time data. AUC (TAU) is the area under the plasma concentration-time curve in one dosing interval.
Time Frame: as for outcome 10
Population: All treated participants with evaluable serum concentration data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Cohort A: Nivolumab 3 mg/kg Q2W | Cohort B: Nivolumab 240 mg Q2W | Cohort C: Nivolumab 360 mg Q3W | Cohort D: Nivolumab 480 mg Q4W
Number analyzed (Participants) | 15 | 20 | 10 | 12
h*ug/mL
  Cycle 1 Day 1 | 8732.232 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 24 | 12112.137 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 24 | 23567.315 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 17 | 49115.208 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 17
  Cycle 3 Day 1: number analyzed (Participants) | 7 | 9 | 0 | 0
  Cycle 3 Day 1 | 30823.993 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 21 | 37794.083 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 22 |  |
  Cycle 5 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 6
  Cycle 5 Day 1 |  |  |  | 100655.626 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 28
  Cycle 6 Day 1: number analyzed (Participants) | 0 | 0 | 7 | 0
  Cycle 6 Day 1 |  |  | 53162.102 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 40 |

14. Secondary Outcome: Ceoinf - Serum Concentration Achieved at the End of Study Drug Infusion
Description: Nivolumab pharmacokinetic parameters are derived from serum concentration versus time data. Ceoinf is the serum concentration achieved at the end of study drug infusion.
Time Frame: End of infusion on Day 1 of Cycle 1, 3, 5, 6
Population: All treated participants with evaluable serum concentration data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Cohort A: Nivolumab 3 mg/kg Q2W | Cohort B: Nivolumab 240 mg Q2W | Cohort C: Nivolumab 360 mg Q3W | Cohort D: Nivolumab 480 mg Q4W
Number analyzed (Participants) | 15 | 18 | 11 | 12
ug/mL
  Cycle 1 Day 1 | 55.020 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 17 | 66.746 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 22 | 93.168 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 23 | 171.494 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 23
  Cycle 3 Day 1: number analyzed (Participants) | 7 | 9 | 0 | 0
  Cycle 3 Day 1 | 122.051 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 17 | 152.058 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 20 |  |
  Cycle 5 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 6
  Cycle 5 Day 1 |  |  |  | 254.704 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 18
  Cycle 6 Day 1: number analyzed (Participants) | 0 | 0 | 7 | 0
  Cycle 6 Day 1 |  |  | 155.811 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 24 |

15. Secondary Outcome: Ctrough - Trough Observed Serum Concentration at the End of Dosing Interval
Description: Nivolumab pharmacokinetic parameters are derived from serum concentration versus time data. Ctrough is the trough observed serum concentration at the end of dosing interval.
Time Frame: Day 1 Cycle 3, 5, 6 (168 hours post dose [Cohort A-B], 336 hours post dose [Cohort C-D])
Population: All treated participants with evaluable serum concentration data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Cohort A: Nivolumab 3 mg/kg Q2W | Cohort B: Nivolumab 240 mg Q2W | Cohort C: Nivolumab 360 mg Q3W | Cohort D: Nivolumab 480 mg Q4W
Number analyzed (Participants) | 7 | 9 | 7 | 6
ug/mL
  Cycle 3 Day 1: number analyzed (Participants) | 7 | 9 | 0 | 0
  Cycle 3 Day 1 | 62.417 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 26 | 62.115 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 39 |  |
  Cycle 5 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 6
  Cycle 5 Day 1 |  |  |  | 92.796 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 39
  Cycle 6 Day 1: number analyzed (Participants) | 0 | 0 | 7 | 0
  Cycle 6 Day 1 |  |  | 61.530 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 35 |

16. Secondary Outcome: Ctau - Concentration at the End of Dosing Interval
Description: Nivolumab pharmacokinetic parameters are derived from serum concentration versus time data. Ctau is the concentration at the end of dosing interval.
Time Frame: as for outcome 10
Population: All treated participants with evaluable serum concentration data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Cohort A: Nivolumab 3 mg/kg Q2W | Cohort B: Nivolumab 240 mg Q2W | Cohort C: Nivolumab 360 mg Q3W | Cohort D: Nivolumab 480 mg Q4W
Number analyzed (Participants) | 13 | 18 | 10 | 12
ug/mL
  Cycle 1 Day 1 | 16.430 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 26 | 20.788 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 30 | 26.143 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 17 | 40.910 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 25
  Cycle 3 Day 1: number analyzed (Participants) | 6 | 8 | 0 | 0
  Cycle 3 Day 1 | 65.286 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 27 | 78.278 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 31 |  |
  Cycle 5 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 5
  Cycle 5 Day 1 |  |  |  | 90.201 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 39
  Cycle 6 Day 1: number analyzed (Participants) | 0 | 0 | 6 | 0
  Cycle 6 Day 1 |  |  | 65.762 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 35 |

17. Secondary Outcome: T-HALFeff - Effective Elimination Half-Life
Description: Nivolumab pharmacokinetic parameters are derived from serum concentration versus time data. T-HALFeff is the effective elimination half-life that explains the degree of observed AUC accumulation calculated based on ratio of an exposure measure at steady state to that after the first dose (exposure measure includes AUC(TAU), Cmax and Ctau).
Time Frame: Day 1 Cycle 3, 5, 6 (pre-dose, 0.5, 4, 8, 24, 48, 96, 168, hours post dose. Cohort C-D includes also 336 hours post dose)
Population: All treated participants with evaluable serum concentration data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Cohort A: Nivolumab 3 mg/kg Q2W | Cohort B: Nivolumab 240 mg Q2W | Cohort C: Nivolumab 360 mg Q3W | Cohort D: Nivolumab 480 mg Q4W
Number analyzed (Participants) | 7 | 9 | 7 | 6
h
  Cycle 3 Day 1: number analyzed (Participants) | 7 | 9 | 0 | 0
  Cycle 3 Day 1 | 551.194 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 24 | 510.262 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 22 |  |
  Cycle 5 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 6
  Cycle 5 Day 1 |  |  |  | 732.44 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 36
  Cycle 6 Day 1: number analyzed (Participants) | 0 | 0 | 7 | 0
  Cycle 6 Day 1 |  |  | 677.642 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 56 |

18. Secondary Outcome: CLT - Total Body Clearance
Description: Nivolumab pharmacokinetic parameters are derived from serum concentration versus time data. CLT is the total body clearance.
Time Frame: as for outcome 17
Population: All treated participants with evaluable serum concentration data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/hr
Arm/Group | Cohort A: Nivolumab 3 mg/kg Q2W | Cohort B: Nivolumab 240 mg Q2W | Cohort C: Nivolumab 360 mg Q3W | Cohort D: Nivolumab 480 mg Q4W
Number analyzed (Participants) | 7 | 9 | 7 | 6
mL/hr
  Cycle 3 Day 1: number analyzed (Participants) | 7 | 9 | 0 | 0
  Cycle 3 Day 1 | 5.732 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 26 | 6.350 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 22 |  |
  Cycle 5 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 6
  Cycle 5 Day 1 |  |  |  | 4.769 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 39
  Cycle 6 Day 1: number analyzed (Participants) | 0 | 0 | 7 | 0
  Cycle 6 Day 1 |  |  | 6.772 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 35 |

19. Secondary Outcome: AI - Accumulation Index (Cmax)
Description: Nivolumab pharmacokinetic parameters are derived from serum concentration versus time data. AI of Cmax refers to the accumulation index calculated based on ratio of an exposure measure of Cmax at steady state to that after the first dose.
Time Frame: as for outcome 17
Population: All treated participants with evaluable serum concentration data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (ug/mL)/(ug/mL)
Arm/Group | Cohort A: Nivolumab 3 mg/kg Q2W | Cohort B: Nivolumab 240 mg Q2W | Cohort C: Nivolumab 360 mg Q3W | Cohort D: Nivolumab 480 mg Q4W
Number analyzed (Participants) | 7 | 9 | 7 | 6
(ug/mL)/(ug/mL)
  Cycle 3 Day 1: number analyzed (Participants) | 7 | 9 | 0 | 0
  Cycle 3 Day 1 | 2.150 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 12 | 2.034 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 15 |  |
  Cycle 5 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 6
  Cycle 5 Day 1 |  |  |  | 1.255 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 29
  Cycle 6 Day 1: number analyzed (Participants) | 0 | 0 | 7 | 0
  Cycle 6 Day 1 |  |  | 1.613 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 17 |

20. Secondary Outcome: AI - Accumulation Index (Ctau)
Description: Nivolumab pharmacokinetic parameters are derived from serum concentration versus time data. AI of Ctau refers to the accumulation index calculated based on ratio of an exposure measure of Ctau at steady state to that after the first dose.
Time Frame: as for outcome 17
Population: All treated participants with evaluable serum concentration data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (ug/mL)/(ug/mL)
Arm/Group | Cohort A: Nivolumab 3 mg/kg Q2W | Cohort B: Nivolumab 240 mg Q2W | Cohort C: Nivolumab 360 mg Q3W | Cohort D: Nivolumab 480 mg Q4W
Number analyzed (Participants) | 6 | 8 | 6 | 5
(ug/mL)/(ug/mL)
  Cycle 3 Day 1: number analyzed (Participants) | 6 | 8 | 0 | 0
  Cycle 3 Day 1 | 3.333 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 25 | 3.215 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 23 |  |
  Cycle 5 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 5
  Cycle 5 Day 1 |  |  |  | 2.053 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 22
  Cycle 6 Day 1: number analyzed (Participants) | 0 | 0 | 6 | 0
  Cycle 6 Day 1 |  |  | 2.675 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 24 |

21. Secondary Outcome: AI - Accumulation Index (AUC)
Description: Nivolumab pharmacokinetic parameters are derived from serum concentration versus time data. AI of AUC refers to the accumulation index calculated based on ratio of an exposure measure of AUC at steady state to that after the first dose.
Time Frame: as for outcome 17
Population: All treated participants with evaluable serum concentration data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (hr*ug/mL)/(hr*ug/mL)
Arm/Group | Cohort A: Nivolumab 3 mg/kg Q2W | Cohort B: Nivolumab 240 mg Q2W | Cohort C: Nivolumab 360 mg Q3W | Cohort D: Nivolumab 480 mg Q4W
Number analyzed (Participants) | 7 | 9 | 7 | 6
(hr*ug/mL)/(hr*ug/mL)
  Cycle 3 Day 1: number analyzed (Participants) | 7 | 9 | 0 | 0
  Cycle 3 Day 1 | 2.942 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 18 | 2.707 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 15 |  |
  Cycle 5 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 6
  Cycle 5 Day 1 |  |  |  | 2.033 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 24
  Cycle 6 Day 1: number analyzed (Participants) | 0 | 0 | 7 | 0
  Cycle 6 Day 1 |  |  | 2.389 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 31 |

22. Primary Outcome: The Number of Participants Experiencing Toxicity Grade 3-4 Laboratory Test Results
Description: The number of participants with Grade 3-4 laboratory results according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0. Note: Grade 4 Toxicities not included in the below table if there were no participants that experienced Grade 4 in that category.
  Grade 3: prolonged recurrence of symptoms following initial improvement; hospitalization indicated for other clinical sequelae [e.g., renal impairment, pulmonary infiltrates].
  Grade 4: Life-threatening; pressor or ventilatory support indicated.
Time Frame: From first dose to 100 days after last dose (up to approximately 28 months)
Population: All treated participants with least one on-treatment measurement of the corresponding laboratory parameter
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Nivolumab 3 mg/kg Q2W | Cohort B: Nivolumab 240 mg Q2W | Cohort C: Nivolumab 360 mg Q3W | Cohort D: Nivolumab 480 mg Q4W
Number analyzed (Participants) | 15 | 20 | 11 | 12
Participants
  HEMOGLOBIN (Grade 3) | 1 | 2 | 0 | 1
  PLATELET COUNT (Grade 3) | 0 | 0 | 0 | 1
  PLATELET COUNT (Grade 4) | 0 | 0 | 0 | 1
  LEUKOCYTES (Grade 3) | 0 | 0 | 2 | 0
  LYMPHOCYTES (ABSOLUTE) (Grade 3) | 0 | 2 | 0 | 1
  ABSOLUTE NEUTROPHIL COUNT (Grade 3) | 0 | 0 | 2 | 0
  ALKALINE PHOSPHATASE (Grade 3) | 2 | 3 | 0 | 0
  ASPARTATE AMINOTRANSFERASE (Grade 3) | 0 | 2 | 0 | 0
  ALANINE AMINOTRANSFERASE (Grade 3) | 0 | 2 | 0 | 0
  BILIRUBIN, TOTAL (Grade 3) | 0 | 1 | 1 | 0
  BILIRUBIN, TOTAL (Grade 4) | 0 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality was assessed from participants first dose to their study completion (up to approximately 28 months). SAEs and Other AEs were assessed from first dose to 100 days following last dose (up to an approximately 14 months, maximum of 28 months)
Arm/Group | Cohort A: Nivolumab 3 mg/kg Q2W | Cohort B: Nivolumab 240 mg Q2W | Cohort C: Nivolumab 360 mg Q3W | Cohort D: Nivolumab 480 mg Q4W
All-Cause Mortality (participants affected / at risk) | 4/15 | 7/20 | 0/11 | 1/12
Serious Adverse Events (participants affected / at risk) | 6/15 | 8/20 | 2/11 | 7/12
Other Adverse Events (participants affected / at risk) | 14/15 | 20/20 | 11/11 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: Nivolumab 3 mg/kg Q2W (N=15) | Cohort B: Nivolumab 240 mg Q2W (N=20) | Cohort C: Nivolumab 360 mg Q3W (N=11) | Cohort D: Nivolumab 480 mg Q4W (N=12)
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0 | 0
Hypothalamo-pituitary disorder (Endocrine disorders) | 0 | 1 | 0 | 0
Optic neuropathy (Eye disorders) | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 0 | 1
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4 | 0 | 1
Brain oedema (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebellar haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0
Paraplegia (Nervous system disorders) | 0 | 0 | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: Nivolumab 3 mg/kg Q2W (N=15) | Cohort B: Nivolumab 240 mg Q2W (N=20) | Cohort C: Nivolumab 360 mg Q3W (N=11) | Cohort D: Nivolumab 480 mg Q4W (N=12)
Anaemia (Blood and lymphatic system disorders) | 3 | 4 | 3 | 4
Granulocytosis (Blood and lymphatic system disorders) | 0 | 0 | 3 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 3 | 3 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 1 | 2 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 3 | 1 | 0
Cardiac discomfort (Cardiac disorders) | 1 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 2 | 1 | 0
Hypothyroidism (Endocrine disorders) | 2 | 6 | 6 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 1
Visual impairment (Eye disorders) | 1 | 1 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Abnormal faeces (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 2 | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 4 | 0 | 3 | 1
Asthenia (General disorders) | 1 | 0 | 0 | 3
Chest discomfort (General disorders) | 0 | 1 | 2 | 0
Chest pain (General disorders) | 2 | 0 | 1 | 0
Chills (General disorders) | 1 | 2 | 0 | 0
Fatigue (General disorders) | 3 | 3 | 1 | 1
Influenza like illness (General disorders) | 0 | 0 | 0 | 1
Malaise (General disorders) | 3 | 6 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 2 | 0 | 0
Pyrexia (General disorders) | 1 | 4 | 4 | 2
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 0
Dacryocystitis (Infections and infestations) | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Otitis media (Infections and infestations) | 1 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 4 | 1 | 3
Upper respiratory tract infection (Infections and infestations) | 1 | 6 | 1 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 3 | 6 | 1 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 6 | 1 | 2
Blood albumin decreased (Investigations) | 0 | 2 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 3 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 2
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 0 | 1
C-reactive protein increased (Investigations) | 0 | 2 | 4 | 0
Granulocyte count increased (Investigations) | 0 | 2 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 3 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 2 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1
Platelet count increased (Investigations) | 0 | 0 | 1 | 0
Protein urine present (Investigations) | 0 | 0 | 2 | 0
Urinary occult blood (Investigations) | 0 | 1 | 1 | 0
Weight decreased (Investigations) | 3 | 1 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 5 | 2 | 1 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 2 | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 5 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 0 | 1
Brain oedema (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 4 | 5 | 0 | 2
Headache (Nervous system disorders) | 3 | 2 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 1
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 3 | 2 | 0 | 0
Poor quality sleep (Psychiatric disorders) | 0 | 0 | 0 | 1
Micturition disorder (Renal and urinary disorders) | 1 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 5 | 3 | 1
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 3 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 1
Laryngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Leukoderma (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Papule (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 5 | 3 | 4 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Telangiectasia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 2 | 0 | 0 | 3
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Phlebitis (Vascular disorders) | 3 | 1 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-15): https://cdn.clinicaltrials.gov/large-docs/86/NCT02593786/Prot_SAP_000.pdf